CLINICAL TRIAL: NCT01579396
Title: The Effects of High-cutoff (HCO) Hemofiltration in the Immediate Postoperative Period on Systemic Inflammatory Response Syndrome (SIRS) and Renal Recovery in Cardiac Surgery Patients With a High Risk for Renal Failure. (HICOSIRS)
Brief Title: High Cut Off Dialysis in Systemic Inflammatory Response Syndrome Patients After Cardiac Surgery
Acronym: HICOSIRS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first patient, due to recruiting problems.
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1486
Record Dates: First submitted 2012-01-18; First posted 2012-04-18 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Systemic Inflammatory Response Syndrome; Acute Kidney Injury
Keywords: septeX; high cut-off; Thoracic Surgery; Renal Replacement Therapy
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Acute Kidney Injury | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- septeX (Experimental): septeX CVVH for 12h after cardiac surgery
  Interventions: Device: septeX
- standard therapy (Other): standard therapy according to local practice
  Interventions: Other: standard therapy

INTERVENTIONS:
Device: septeX — 12 h septeX CVVH treatment after cardiac surgery
  Other Names: high cut off
  Arms: septeX
Other: standard therapy — standard therapy either pharmacological and /or continuous renal replacement therapy (CRRT)
  Arms: standard therapy

SUMMARY:
A high cut off dialyzer (septeX) is tested in patients after cardio-thoracic surgery with incidence of "systemic inflammatory response syndrome" (SIRS) and associated increased risk for acute kidney injury (AKI). Hypothesis: The high cut off dialyzer (septeX) can increase the postoperative IL-6/Il-10 ratio.

DETAILED DESCRIPTION:
Cardiac surgery associated systemic inflammatory response syndrome (SIRS) plays an important pathophysiological role in the development of AKI in patients after cardiothoracic surgery.

Previous studies have shown that the elimination of inflammatory mediators can be either achieved by Continuous Venous Venous Hemodialysis(CVVHD) or Continuous Venous Venous Hemofiltration (CVVH) by using a high-cutoff (HCO) membrane with a cut-off 45kD. Data from patients treated with HCO-CVVHD during septic shock show a reduction in systemic cytokines and improved hemodynamics.

No data about the effects of early HCO-CVVH in cardiac surgery patients with a high risk of Cardiac Surgery associated AKI and consequently a high rate of postoperative renal replacement therapy (RRT) are available.

It is of note that patients with Euroscore > 6 are on high risk to develop SIRS associated AKI.

No pharmacological anti-inflammatory approach has convincingly shown to prevent renal dysfunction in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for complex / prolonged cardiac surgery (i.e.combined CABG+ valve surgery, Redo surgery) with an anticipated CPB time > 120 min
* CKD with an e GFR < 50ml/min/m2
* Euroscore > 6

Exclusion Criteria:

* End stage CKD (dialysis dependent) renal failure before surgery
* Radiocontrast exposure within 24 hours before surgery
* Active endocarditic with antibiotic treatment
* pulmonary disease with chronic hypoxia
* Clinically significant liver dysfunction (bilirubin > 1.8mg/dl (30µmol/L))
* Known HIV, HCV infection
* Alcoholism
* Active uncontrolled infection
* Pregnancy or lactation
* Inability to give informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
IL6/IL10 ratio | Change from Baseline in IL6/IL10 ratio at 48h post cardiac surgery and last day at hospital (expected average of 2 weeks after cardiac surgery)
  To test, if immediate postoperative HCO-CVVH reduces systemic inflammation (determined as the ratio between Il-6 / Il-10) in patients with a high risk for CSA-AKI in comparison with a treatment without early RRT. To calibrate for differences in baseline cytokine levels and with respect to the high variability of cytokines in the postoperative period the area-under-the-curve (AUC) of the postoperative increase in the IL-6/Il-10 ratio until 48h will be used.

SECONDARY OUTCOMES:
determination of immediate postoperative HCO-CVVH improvement | 6 month post cardiac surgery
  * Short- and medium term recovery of renal function
  * time to extubation
  * cardiac function
  * need for vasoactive and inotropic drugs
  * duration of treatment in a high-dependency unit
Laboratory assessments | 48h after cardiac surgery and last day at hospital (expected average 2 weeks)
  * GDF-15
  * urinary fatty acid binding protein (U-FABP)
  * association of Human placental growth factor (PIGF) and Soluble fms-like tyrosine kinase (S-flt-1)
adverse effects | 48h after cardiac surgery
  To determine, if HCO - CVVH has adverse effects in comparison with no immediate RRT.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Heringlake, Prof. Dr., Principal Investigator — Universitaet zu Luebeck
Locations (1):
- Klinik für Anaesthesiologie UKSH Luebeck, Lübeck, Schleswig-Holstein, Germany